CLINICAL TRIAL: NCT06636578
Title: Dexmedetomidine Ropivacaine Versus Plain Ropivacaine in Bilateral Pectoralis Nerve (PECS) Block for Fast Tracking and Postoperative Analgesia in Open Heart Surgery Through Midline Sternotomy. A Randomized Clinical Trial
Brief Title: Dexmedetomidine Ropivacaine Versus Plain Ropivacaine in Bilateral Pectoralis Nerve (PECS) Block
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate Professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R 611
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Analgesia
Keywords: PECS block; analgesia after median sternotomy
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Ropivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (DR) (Active Comparator): will receive 30 ml of 0.25% ropivacaine + dexmedetomidine 0.5 μg/kg for each side.
  Interventions: Drug: dexmedetomidine; Drug: ropivacaine
- Group (R) (Active Comparator): will receive 30 ml of 0.25% of plain ropivacaine for each side.
  Interventions: Drug: ropivacaine
- Group (C) (Sham Comparator): the control group will not receive any regional anesthesia and only will receive fentanyl 1μg/kg/hr.
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: dexmedetomidine — will receive 30 ml of 0.25% of ropivacaine + dexmedetomidine 0.5 μg/kg for each side.
  Other Names: precedex
  Arms: Group (DR)
Drug: ropivacaine — will receive 30 ml of 0.25% of plain ropivacaine for each side.
  Other Names: plain ropivacaine
  Arms: Group (DR); Group (R)
Drug: fentanyl — will not receive any regional anesthesia and only will receive I.V. fentanyl 1μg/kg/hr.
  Arms: Group (C)

SUMMARY:
In 2012 Blanco et al. [1] described the ultrasound technique for Pectoral nerve (PECS) block as a new, less invasive regional analgesic technique for breast surgeries.

PECS block includes PECS I and PECS II (modified PECS I) interfascial blocks. Since that time, PECS block has been used successfully with good results for a wide variety of surgeries on the chest wall such as radical mastectomies, breast-conserving surgeries, breast implant placement, automated implantable cardioverter-defibrillator (AICD)/pacemaker placement, intercostal drainage tube placement, and rib fractures. In this study, the investigators hypothesized that adding dexmedetomidine as an adjuvant to ropivacaine can result in the prolongation of the duration of anesthesia with improvement of the quality of postoperative analgesia of bilateral PECS block for patients undergoing cardiac surgery via midline sternotomy compared with using only plain ropivacaine.

DETAILED DESCRIPTION:
This study will be performed at the FAYOUM University Hospital after approval from the local Institutional Ethics Committee and the local Institutional Review Board. It will be a double-blind randomized controlled study. The eligible patients will sign a detailed informed consent form before recruitment and randomization.

After confirming hemodynamic stability, satisfactory blood gasses, electrolytes, normalized activated coagulation time (ACT < 120 s), and minimal drain output, bilateral PECS block will be performed guided by a linear ultrasound transducer (12 MHz). 5

The block will be performed in a supine position with the arm slightly abducted. Under complete aseptic precautions, and using a 20 gauge 5 cm needle. The ultrasound probe will be placed at the midclavicular level inferolaterally to locate the axillary artery and vein and then moved laterally toward the axilla until pectoralis major, pectoralis minor, and serratus anterior muscles were identified at the level of the fourth rib.

The needle will be inserted in the plane concerning the ultrasound probe. A volume of 20 ml of local anesthetic solution will be deposited in the fascial plane between pectoralis minor and serratus anterior muscle, followed by withdrawal of the needle to the fascial plane between pectoralis major and pectoralis minor muscle, where a volume of 10 ml will be deposited. The block will be performed similarly on both sides. It will be noted that the total dose of local anesthetic is not to exceed the toxic dose of ropivacaine (3 mg/kg). Patients then will be transferred intubated to the Surgical ICU (SICU), and standard monitoring will be continued until patients are fully awake, patients will be extubated once they fulfilled the extubation criteria.

Sample Size ( number of participants included ) 90 patients

Methodology in detail:

All patients will receive a slandered anesthesia technique. The main goal of the anesthesia technique will be to ensure a rapid return of consciousness and protective reflexes, with minimal residual sedative effects, and importantly, it should facilitate early ambulation. Continuous infusion of fentanyl, midazolam, and rocuronium as total intravenous anesthesia (TIVA).

At the end of the surgery, TIVA will be stopped, and paracetamol 1 gm IV infusion over 15 min will be administered with closure of the sternum.

After dressing, Patients will be randomly allocated into three groups:

Group (C) control group (n = 30): will not receive any regional anesthesia and only will receive fentanyl 1μg/kg/hr.

For the other two groups, regional anesthesia will be used, and every patient in these two groups will receive 20 ml of ropivacaine 0.25% will be used by the surgeon for infiltration in the surgical incision site and in the skin around the mediastinal drains. In addition, every patient in these two groups will receive bilateral ultrasound-guided PECS block as follows:

Group (R) (n = 30): will receive 30 ml of 0.25% of plain ropivacaine for each side.

Group (DR) (n = 30): will receive 30 ml of 0.25% of ropivacaine + dexmedetomidine 0.5 μg/kg for each side.

Measured data:

1. pain assessment will be done using the VAS scoring system (On a pain scale [0-10] at rest and during cough by an intensivist blinded to the study groups at 0 h (at extubation) and thereafter at 3, 6, 12, 18, and 24 h intervals. Pain will be classified into mild, moderate, and severe for analysis (mild VAS 0-4, moderate VAS 5-7, and severe VAS >8).
2. Duration of mechanical ventilation.
3. total dose of fentanyl used for breakthrough pain.
4. incidence of any complications.
5. duration of ICU stay.
6. Patient's satisfaction level will be assessed with a Likert five-item scoring system

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 65 years,
* Ejection fraction (EF) > 35%,
* Elective isolated CABG, or Valve surgery

Exclusion Criteria:

* Poor left ventricular function with intra-aortic balloon pump support,
* Recent myocardial infarction (last seven days),
* Combined procedure (i.e., CABG + other heart/vascular procedure),
* Emergency surgery, or Redo cases,
* Hepatic or renal failure, creatinine >1.5,
* Patients with hemodynamic instability, preexisting infection at the site of block, allergy to local anesthetics, psychiatric illness, and patients with prolonged postoperative ventilatory course were excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-08 (Estimated)

PRIMARY OUTCOMES:
pain assessment will be done using VAS scoring system | The first 24 hours postoperative
  (In a pain scale [0-10] at rest and during cough by an intensivist blinded to the study groups at 0 h (at extubation) and thereafter at 3, 6, 12, 18, and 24 h intervals. Pain will be classified into mild, moderate, and severe for analysis (mild VAS 0-4, moderate VAS 5-7, and severe VAS >8)
Total opioid consumption | from the time of ICU admission hour 1 up to hour 24
  the amount of opioid (mostly used is fentanyl amp. in equivalent doses ) that has been used for 24 hours after admission in ICU

CONTACTS AND LOCATIONS:
Overall Officials: mohamed hamed, M.D, Principal Investigator — Fayoum University
Locations (2):
- Egypt (2):
  - Fayoum University Hospital, Al Fayyum
  - Mohamed Hamed, Al Fayyum

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sertcakacilar G, Tire Y, Kelava M, Nair HK, Lawin-O'Brien ROC, Turan A, Ruetzler K. Regional anesthesia for thoracic surgery: a narrative review of indications and clinical considerations. J Thorac Dis. 2022 Dec;14(12):5012-5028. doi: 10.21037/jtd-22-599. PMID 36647492
- [Background] Kumar KN, Kalyane RN, Singh NG, Nagaraja PS, Krishna M, Babu B, Varadaraju R, Sathish N, Manjunatha N. Efficacy of bilateral pectoralis nerve block for ultrafast tracking and postoperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):333-338. doi: 10.4103/aca.ACA_15_18. PMID 30052231
- [Background] Yalamuri S, Klinger RY, Bullock WM, Glower DD, Bottiger BA, Gadsden JC. Pectoral Fascial (PECS) I and II Blocks as Rescue Analgesia in a Patient Undergoing Minimally Invasive Cardiac Surgery. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):764-766. doi: 10.1097/AAP.0000000000000661. PMID 29016551